CLINICAL TRIAL: NCT04040582
Title: Psychedelics and Wellness Study (PAWS): An Online Anonymous Survey Investigating the Interrelationship Between Past Psychedelic Use and Its Impact on Levels of Wellness
Brief Title: Psychedelics and Wellness Study (PAWS)
Acronym: PAWS
Status: Completed | Type: Observational
Sponsor: WILD 5 Wellness (Other)
Responsible Party: Principal Investigator, Saundra Jain, MA, PsyD, LPC, Psychotherapist, WILD 5 Wellness
Other Study IDs: WILD 5 Wellness
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Depression, Anxiety, PTSD
Keywords: Psychedelics, Wellness
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Psychedelics and Wellness Study (PAWS), is an anonymous online survey investigating the interrelationship between psychedelics and wellness. The study population is adults ages 18 and older that have taken a psychedelic at least once. The maximum sample size is 5,000 survey respondents. It is expected that this anonymous online survey will support the hypothesis that there is a robust interrelationship between past psychedelic use and its impact on wellness.

DETAILED DESCRIPTION:
Following a four-decade moratorium, the therapeutic use of psychedelics has once more captured the collective attention of the medical community and the public at large. Now, at the forefront of a renaissance in psychedelic research, this study is investigating the interrelationship of psychedelics and mental wellness - a state of well-being in which the individual realizes his or her own abilities, can cope with the normal stresses of life, can work productively and fruitfully, and is able to make a contribution to his or her community. This work will be unique in that it will collect both objective and subjective data to assess the interrelationship between psychedelic and wellness. It will lend support to the growing body of research in the use of psychedelics for both mental health conditions and the pursuit of overall mental wellness.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 and older that have taken a psychedelic at least once.

Exclusion Criteria:

* Individuals less than 18 years old and have previously never taken a psychedelic substance.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults ages 18 and older that have taken a psychedelic at least once.
Sampling Method: Non-Probability Sample
Enrollment: 3234 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Through study completion, an average of 1 year
  The PHQ-9 is a nine-item depression self-report questionnaire for screening and measurement of severity of major depression. Scores range from 0-27 (Lower scores = Less depression).
Change in Generalized Anxiety Disorder-7 (GAD-7) | Through study completion, an average of 1 year
  The GAD-7 is a seven-item self-report questionnaire for screening and measurement of severity of generalized anxiety disorder. Scores range from 0-21 (Lower scores = Less anxiety).
Change in HERO Wellness Scale | Through study completion, an average of 1 year
  The HERO Wellness Scale is a brief 5-item scale designed to measure four wellness traits plus perceived mental wellness. Scores range from 0-50 (Lower scores = Lower levels of mental wellness).

CONTACTS AND LOCATIONS:
Overall Officials: Saundra Jain, PsyD, LPC, Principal Investigator — WILD 5 Wellness
Locations (1):
- WILD 5 Wellness, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data that will be shared with other researchers will not be identified by participant; it will only be shared in aggregate form.

REFERENCES:
- [Derived] Herrmann Z, Levin AW, Cole SP, Slabaugh S, Barnett B, Penn A, Jain R, Raison C, Rajanna B, Jain S. Psychedelic Use Among Psychiatric Medication Prescribers: Effects on Well-Being, Depression, Anxiety, and Associations with Patterns of Use, Reported Harms, and Transformative Mental States. Psychedelic Med (New Rochelle). 2023 Sep 13;1(3):139-149. doi: 10.1089/psymed.2023.0030. eCollection 2023 Sep. PMID 40046570